CLINICAL TRIAL: NCT00808990
Title: Probiotics and Non Alcoholic Steatohepatitis (NASH)
Brief Title: The Effect of Probiotics on Non Alcoholic Fatty Liver Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Time table was unfulfilled due to incompetent research coordinator. Inaccurate results and No conclusions can be withdrawn
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, weiss hemda, Dr., Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMC085077CTIL; RMC local ID 5077
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Liver Disease
Keywords: Non Alcoholic Fatty Liver Disease; Non Alcoholic SteatoHepatitis; Small bowel bacterial overgrowth; Probiotics; Patients with Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSA and NAFLD patients using CPAP (Experimental): OSA and NAFLD patients using CPAP being followed for 6 months.
  Interventions: Dietary Supplement: BioFemale
- control (No Intervention): OSA and NAFLD patients not using CPAP being followed for 6 months.

INTERVENTIONS:
Dietary Supplement: BioFemale — BioFemale 6 months.
  Arms: OSA and NAFLD patients using CPAP

SUMMARY:
Nonalcoholic Fatty Liver Disease (NAFLD) has been suggested to be the most common cause of chronic liver disease in the general population in the Western World. In advanced stages of NAFLD, steatohepatitis (NASH) develops characterized by: steatosis, inflammation, and fibrosis progressing to cirrhosis in some patients. The knowledge of the role of small intestinal bacterial overgrowth (SIBO) in the pathogenesis of NASH has led to the proposal of probiotics as a therapeutic strategy for this disorder.

DETAILED DESCRIPTION:
Probiotics may interfere with the development of NASH by several mechanisms. Data from an uncontrolled clinical trial in NASH patients show promising results, with improvement of liver enzymes in treated patients.

RESEARCH GOALS:

A. To assess the degree of SIBO in NAFLD patients vs. healthy controls. B. To evaluate the effect of probiotics vs. placebo on SIBO in NAFLD patients. C. To evaluate the effect of probiotics vs. placebo on disease severity (inflammation, steatosis, and fibrosis) in NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

* Controls- healthy volunteers, male and female, above 18 years.
* NAFLD group - patients with histological proven NAFLD, male and female, above 18 years.

Exclusion Criteria:

* Controls

  * those who will be found to have fatty liver in abdominal ultra sound
  * any participant who will take antibiotics for any indication for more than 1 week during the study period or before recruitment to the study
  * any participant who had lost more than 10% of baseline body weight during the study period.
* NAFLD group

  * those who will be found to have any concomitant liver disease (i.e., HBV/HCV/HIV/EBV/CMV infection
  * autoimmune hepatitis
  * metabolic liver disease: Wilson's disease, cholestatic liver disease: PBC/PSC, etc.)
  * any participant who will take antibiotics for any indication for more than 1 week during the study period or before recruitment to the study
  * any participant who had lost more than 10% of baseline body weight during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
SIBO in NASH patients in both treated groups (probiotics treated versus placebo treated) will be evaluated by lactulose breath test | Recruitment period of 6 months and 6 months of treatment after each recruitment
Lactulose breath test | Measurement at recruitment (0) and at the end of treatment period (6 mo)

SECONDARY OUTCOMES:
FIBROMAX tests will assess severity of NAFLD in patients' group prior to treatment and post treatment | At recruitment to the study (0) and at the end of treatment (6 mo)
Fibromax test for the evaluation of NAFLD severity | At the recruitment (0) and at the end of treatment (6 mo)

CONTACTS AND LOCATIONS:
Overall Officials: Hemda Weiss, M.D., Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Li Z, Yang S, Lin H, Huang J, Watkins PA, Moser AB, Desimone C, Song XY, Diehl AM. Probiotics and antibodies to TNF inhibit inflammatory activity and improve nonalcoholic fatty liver disease. Hepatology. 2003 Feb;37(2):343-50. doi: 10.1053/jhep.2003.50048. PMID 12540784
- [Background] Loguercio C, De Simone T, Federico A, Terracciano F, Tuccillo C, Di Chicco M, Carteni M. Gut-liver axis: a new point of attack to treat chronic liver damage? Am J Gastroenterol. 2002 Aug;97(8):2144-6. doi: 10.1111/j.1572-0241.2002.05942.x. No abstract available. PMID 12190198
- [Background] Khoshini R, Dai SC, Lezcano S, Pimentel M. A systematic review of diagnostic tests for small intestinal bacterial overgrowth. Dig Dis Sci. 2008 Jun;53(6):1443-54. doi: 10.1007/s10620-007-0065-1. PMID 17990113
- [Background] Nair S, Cope K, Risby TH, Diehl AM. Obesity and female gender increase breath ethanol concentration: potential implications for the pathogenesis of nonalcoholic steatohepatitis. Am J Gastroenterol. 2001 Apr;96(4):1200-4. doi: 10.1111/j.1572-0241.2001.03702.x. PMID 11316170
- [Background] Yang SQ, Lin HZ, Lane MD, Clemens M, Diehl AM. Obesity increases sensitivity to endotoxin liver injury: implications for the pathogenesis of steatohepatitis. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2557-62. doi: 10.1073/pnas.94.6.2557. PMID 9122234
- [Background] Chitturi S, Farrell GC. Etiopathogenesis of nonalcoholic steatohepatitis. Semin Liver Dis. 2001;21(1):27-41. doi: 10.1055/s-2001-12927. PMID 11296694
- [Background] Wigg AJ, Roberts-Thomson IC, Dymock RB, McCarthy PJ, Grose RH, Cummins AG. The role of small intestinal bacterial overgrowth, intestinal permeability, endotoxaemia, and tumour necrosis factor alpha in the pathogenesis of non-alcoholic steatohepatitis. Gut. 2001 Feb;48(2):206-11. doi: 10.1136/gut.48.2.206. PMID 11156641
- [Background] Solga SF, Buckley G, Clark JM, Horska A, Diehl AM. The effect of a probiotic on hepatic steatosis. J Clin Gastroenterol. 2008 Nov-Dec;42(10):1117-9. doi: 10.1097/MCG.0b013e31816d920c. No abstract available. PMID 18936646